CLINICAL TRIAL: NCT01087970
Title: Phase 2 Study of Pemetrexed in Combination With Carboplatin or Cisplatin and Cetuximab in Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: A Study for Participants With Recurrent or Metastatic Squamous Cell Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13491; H3E-MC-S132 (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-03-15; First posted 2010-03-16 (Estimated); Results first posted 2014-05-19 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-04

CONDITIONS: Head and Neck Neoplasms
Keywords: Pharynx; Larynx; Nose; Parathyroid
MeSH Terms: conditions — Head and Neck Neoplasms; Laryngeal Diseases | interventions — Pemetrexed; Cetuximab; Carboplatin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Triplet Combination Therapy (Experimental): Cycle 1:
  Week 1 - Cetuximab 400 milligrams/square meter (mg/m²) on Day 1; Pemetrexed 500 mg/m² on Day 1; Carboplatin area under curve (AUC) 5 on Day 1 or Cisplatin 75 mg/m² on Day 1
  Week 2 - Cetuximab 250 mg/m² on Day 1
  Week 3 - Cetuximab 250 mg/m² on Day 1
  Cycle 2-6:
  Week 1 - Cetuximab 250 mg/m² on Day 1; Pemetrexed 500 mg/m² on Day 1; Carboplatin AUC 5 on Day 1 or Cisplatin 75 mg/m² on Day 1
  Week 2 - Cetuximab 250 mg/m² on Day 1
  Week 3 - Cetuximab 250 mg/m² on Day 1
  Following Cycle 6, Cetuximab Monotherapy: 250 mg/m² intravenously weekly on Day 1
  Interventions: Drug: Pemetrexed; Drug: Cetuximab; Drug: Carboplatin; Drug: Cisplatin

INTERVENTIONS:
Drug: Pemetrexed — Administered intravenously, for maximum of 6 cycles.
  Other Names: Alimta; LY231514
Drug: Cetuximab — Administered intravenously in combination therapy, for a maximum of 6 cycles.
  After the completion of 6 cycles, participants who have not experienced disease progression will continue on cetuximab monotherapy until disease progression.
  Other Names: Erbitux
Drug: Carboplatin — Administered intravenously, for a maximum of 6 cycles
Drug: Cisplatin — Administered intravenously, for a maximum of 6 cycles

SUMMARY:
The purpose of this study is to look for an improvement in progression free survival with the combination of pemetrexed, carboplatin (or cisplatin) and cetuximab in participants with recurrent or metastatic squamous cell carcinoma of the head and neck.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of squamous cell head and neck cancer (HNC)

  * Recurrent disease (locally advanced or metastatic) that is not amenable to local therapy, (i) with at least 6 months since completion of systemic therapy (chemotherapy or biological anticancer therapy), and (ii) with no more than 1 prior multimodal therapy (such as concurrent chemoradiation with or without sequential chemotherapy) for locally advanced HNC tumor, and (iii) with no prior systemic therapy (chemotherapy or biological anticancer therapy) for metastatic disease; OR
  * Newly diagnosed distant metastatic disease (Stage IVc)
* Prior therapies:

  * Radiation therapy must be completed at least 4 weeks before study enrollment. For palliative therapy, prior radiation therapy allowed <25% of the bone marrow and prior radiation to the whole pelvis is not allowed. Participants must have recovered from the acute toxic effects of the treatment prior to study enrollment.
  * Surgery (excluding prior diagnostic biopsy) must be completed at least 4 weeks before study enrollment. Participants must have fully recovered from any acute effects of surgery prior to study enrollment.
* An estimated life expectancy of at least 12 weeks.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Biological tissue available for biomarker analysis on tumor tissue.
* Disease status must be measurable as defined by Response Evaluation Criteria in Solid Tumors (RECIST). The index lesion must not be in a prior irradiated area. Positron emission tomography (PET) scans and ultrasounds may not be used for lesion measurements.
* Participant compliance and geographic proximity that allow for adequate follow-up.
* Adequate organ function as defined by the following:

  * Bone marrow reserve: absolute neutrophil (segmented and bands) count (ANC) greater than or equal to 1.5 × 10⁹/liter (L), platelets greater than or equal to 100 × 10⁹/L, and hemoglobin greater than or equal to 9 grams/deciliter (g/dL).
  * Hepatic: bilirubin less than or equal to 1.5 × the upper limit of normal (ULN); alkaline phosphatase (ALP), aspartate aminotransferase (AST), and alanine aminotransferase (ALT) less than or equal to 3.0 × ULN (ALP, AST, and ALT less than or equal to 5.0 × ULN is acceptable if the liver has tumor involvement).
  * Renal: calculated creatinine clearance (CrCl) greater than or equal to 45 milliliters/minute (mL/min).
* For women: Must be surgically sterile, postmenopausal, or compliant with a medically approved contraceptive regimen during and for 6 months after the treatment period; must have a negative serum or urine pregnancy test within 7 days before study enrollment, and must not be breast-feeding. For men: Must be surgically sterile or compliant with a contraceptive regimen during and for 6 months after the treatment period.

Exclusion Criteria:

* Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry.
* Are receiving concurrent chronic systemic immune therapy, or chemotherapy for a disease other than cancer.
* Concurrent administration of any other antitumor therapy.
* Known prior allergic/hypersensitivity reaction to any of the components of the study treatment.
* Serious concomitant systemic disorder (for example, active infection) or psychiatric disorder that, in the opinion of the investigator, would compromise the participant's ability to complete the study.
* Have serious cardiac disease, such as symptomatic angina, unstable angina, or the history of myocardial infarction in the previous 12 months.
* Second primary malignancy that is clinically detectable at the time of consideration for study enrollment.
* Have had another primary malignancy other than HNC, unless that prior malignancy was treated at least 2 years previously with no evidence of recurrence. Exception: Participants with a history of in situ carcinoma of the cervix, nonmelanoma skin cancer, or low-grade (Gleason score less than or equal to 6) localized prostate cancer will be eligible even if diagnosed and treated less than 2 years previously.
* Nasopharyngeal, paranasal sinus, lip, or salivary gland cancer.
* Presence of clinically significant (by physical exam) third-space fluid collections; for example, ascites or pleural effusions that cannot be controlled by drainage or other procedures prior to study entry.
* Have peripheral neuropathy of Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 or higher.
* Have central nervous system (CNS) metastases (unless the participant has completed successful local therapy for CNS metastases and has been off corticosteroids for at least 4 weeks before starting study therapy). Brain imaging is required in symptomatic participants to rule out brain metastases, but is not required in asymptomatic participants.
* Inability to interrupt aspirin or other nonsteroidal anti-inflammatory agents, other than an aspirin dose less than or equal to 1.3 grams per day, for a 5-day period (8-day period for long-acting agents, such as piroxicam).
* Unable or unwilling to take folic acid, vitamin B12, or prophylactic corticosteroids.
* Recent (within 30 days before enrollment) or concurrent yellow fever vaccination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2010-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (21):
- United States (21):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jonesboro, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Waterbury, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Myers, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marietta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Savannah, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valdosta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Scarborough, Maine
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Detroit, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Louis Park, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Billings, Montana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buffalo, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., The Bronx, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbia, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sioux Falls, South Dakota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chattanooga, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Richmond, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Cetuximab + Pemetrexed + Carboplatin/Cisplatin: Cetuximab loading dose of 400 milligrams/square meter (mg/m²) administered intravenously on Day 1 of Cycle 1; subsequently 250 mg/m² intravenously weekly.
  Pemetrexed 500 mg/m² administered intravenously on Day 1 of every 21-day cycle, 1 hour after cetuximab.
  Carboplatin area under curve (AUC) 5 or cisplatin 75 mg/m² administered intravenously on Day 1 of every 21-day cycle, 30 minutes after pemetrexed.
  Maximum 6 cycles. Participants who did not experience disease progression after 6 cycles continued on cetuximab (250 mg/m² intravenously weekly) monotherapy until disease progression.
Period: Overall Study
Arm/Group | Cetuximab + Pemetrexed + Carboplatin/Cisplatin
Started | 69
Received ≥1 Dose of Any Study Drug | 69
Completed 6 Cycles | 69
Efficacy Population | 58 (All treated participants excluding those from a noncompliant study site.)
Received Carboplatin | 63
Completed | 67
Not Completed | 2
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least 1 dose of study drug.
Groups:
- Cetuximab + Pemetrexed + Carboplatin/Cisplatin: Cetuximab loading dose of 400 mg/m² administered intravenously on Day 1 of Cycle 1; subsequently 250 mg/m² intravenously weekly.
  Pemetrexed 500 mg/m² administered intravenously on Day 1 of every 21-day cycle, 1 hour after cetuximab.
  Carboplatin AUC 5 or cisplatin 75 mg/m² administered intravenously on Day 1 of every 21-day cycle, 30 minutes after pemetrexed.
  Maximum 6 cycles. Participants who did not experience disease progression after 6 cycles continued on cetuximab (250 mg/m² intravenously weekly) monotherapy until disease progression.
Arm/Group | Cetuximab + Pemetrexed + Carboplatin/Cisplatin
Number analyzed (Participants) | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 63
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 11
  White | 56
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 69
European-Quality of Life-5 Dimension Instrument-3 Levels (EQ-5D-3L) [Mean (Standard Deviation); unit: units on a scale] — Participants assessed health-related QoL in 5 D (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) as no problems/some or moderate problems/extreme problems. A regression equation defines a utility value for these health states to generate an index score from -0.594 (severe problems in all 5 D) to 1 (no problem in all 5 D) where 1=best possible health state. EQ-5D VAS rates participant's current health-related QoL on the day of questionnaire administration and is captured on a scale of 0 (worst imaginable health state) to 100 (best imaginable health state).
  units on a scale
    Index Score (n=47) | 0.721 (0.248)
    Visual Analog Scale (VAS) Score (n=47) | 66.106 (20.658)
Performance Status Scale for Head and Neck Cancer (PSS-HNC) [Mean (Standard Deviation); unit: units on a scale] — Clinician measured speaking and eating disabilities of HNC participants that consists 3 subscales: normalcy of diet (NOD) measures ability of eating a normal diet, scale from 0 (non-oral feeding) to 100 (unrestricted diet); understandability of speech (UOS) measures the degree a clinician was able to understand participant's speech, scale from 0 (never understandable) to 100 (always understandable); eating in public (EIP) is based on clinician's question to the participant, scale from 0 (always eats alone) to 100 (no restriction of place, food, or companion).
  units on a scale
    NOD (n=57) | 56.32 (37.87)
    UOS (n=57) | 78.51 (32.20)
    EIP (n=57) | 71.93 (34.42)

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the duration from the date of enrollment to the first date of documented objective progressive disease (PD) or death from any cause. PD was determined using Response Evaluation Criteria In Solid Tumors (RECIST) criteria version 1.0. PD is ≥20% increase in sum of longest diameter of target lesions or the appearance of new lesions. For participants who were not known to have died or to have had objective PD at the time of the data inclusion cutoff, PFS was censored at their last objective progression-free disease assessment prior to the cutoff date or the date of initiation of subsequent systemic anticancer therapy.
Time Frame: From enrollment to measured progressive disease up to 15.3 months (tumor assessments performed every other cycle during study treatment, and then every 6 weeks during follow-up)
Population: All treated participants excluding those from a noncompliant study site. The number of participants censored was 9.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Cetuximab + Pemetrexed + Carboplatin/Cisplatin: Cetuximab loading dose of 400 mg/m² administered intravenously on Day 1 of Cycle 1; subsequently 250 mg/m² administered intravenously weekly.
  Pemetrexed 500 mg/m² administered intravenously on Day 1 of every 21-day cycle, 1 hour after cetuximab.
  Carboplatin AUC 5 or cisplatin 75 mg/m² administered intravenously on Day 1 of every 21-day cycle, 30 minutes after pemetrexed.
  Maximum 6 cycles. Participants who did not experience disease progression after 6 cycles continued on cetuximab (250 mg/m² intravenously weekly) monotherapy until disease progression.
Arm/Group | Cetuximab + Pemetrexed + Carboplatin/Cisplatin
Number analyzed (Participants) | 58
months | 5.1 [3.9 to 6.0]

2. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the duration from the date of enrollment to the date of death from any cause. For participants who were alive at the time of the data inclusion cutoff, OS was censored at the date of last contact prior to that cut-off date.
Time Frame: From enrollment to the date of death from any cause up to 26.4 months (assessment completed during trial period at least every 3 months)
Population: All treated participants excluding those from a noncompliant study site. The number of participants censored was 22.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab + Pemetrexed + Carboplatin/Cisplatin
Number analyzed (Participants) | 58
months | 11.1 [7.6 to 14.8]

3. Secondary Outcome: Percentage of Participants Having a Confirmed Partial Response (PR) or Complete Response (CR)
Description: PR or CR is classified by the investigators according to RECIST criteria version 1.0. PR is a ≥30% decrease in sum of longest diameter of target lesions without new lesion and progression of non-target lesions; CR is the disappearance of all target and non-target lesions. Percentage of participants having a PR or CR is calculated as a total number of participants with PR or CR from enrollment until disease progression or recurrence divided by the total number of participants treated, then multiplied by 100.
Time Frame: From enrollment to objectively determined progressive disease up to 15.3 months (tumor assessments performed every other cycle during study treatment until progressive disease)
Population: All treated participants excluding those from a noncompliant study site.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab + Pemetrexed + Carboplatin/Cisplatin
Number analyzed (Participants) | 58
percentage of participants | 25.9 [15.3 to 39.0]

4. Secondary Outcome: Change From Baseline in Participant-Reported European-Quality of Life-5 Dimension Instrument-3 Levels (EQ-5D-3L)
Description: EQ-5D-3L is a descriptive system of health-related quality of life states consisting of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and each of which has 3 levels of severity (no problems/some or moderate problems/extreme problems) within a particular EQ-5D dimension. A regression equation defines a utility value for these health states to generate an index score. The possible values for index score range from -0.594 (severe problems in all 5 dimensions) to 1 (no problem in all dimensions) on a scale where 1 represents the best possible health state. The EQ-5D Visual Analog Scale (VAS) is used to record a participant's rating for his/her current health-related quality of life state on the day of questionnaire administration and is captured on a scale of 0 (worst imaginable health state) to 100 (best imaginable health state).
Time Frame: Baseline, Day 1 of Cycles 2, 4, 6, cetuximab monotherapy Cycles 2 and 4 (21-day cycle)
Population: All treated participants who completed the EQ-5D-3L and VAS at baseline and in Cycles 2, 4, 6, cetuximab monotherapy Cycles 2 and 4. Exclude those from a noncompliant study site.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cetuximab + Pemetrexed + Carboplatin/Cisplatin
Number analyzed (Participants) | 43
units on a scale
  Change in Index Score at Cycle 2 (n=43) | 0.038 (0.233)
  Change in Index Score at Cycle 4 (n=29) | 0.070 (0.147)
  Change in Index Score at Cycle 6 (n=24) | -0.063 (0.249)
  Change in Index Score at monotherapy Cycle2 (n=14) | 0.016 (0.098)
  Change in Index Score at monotherapy Cycle 4 (n=7) | 0.059 (0.080)
  Change in VAS Score at Cycle 2 (n=41) | 3.854 (21.600)
  Change in VAS Score at Cycle 4 (n=28) | 2.107 (24.894)
  Change in VAS Score at Cycle 6 (n=21) | 0.333 (16.716)
  Change in VAS Score at monotherapy Cycle 2 (n=14) | -1.500 (16.919)
  Change in VAS Score at monotherapy Cycle 4 (n=7) | 0.571 (13.377)

5. Secondary Outcome: Change From Baseline in Performance Status Scale for Head and Neck Cancer (PSS-HNC)
Description: PSS-HNC is a clinician-rated instrument designed to measure speaking and eating disabilities of participants with head and neck cancer and consists of 3 subscales: normalcy of diet (NOD) subscale measures the ability of the participants to eat a normal diet, subscale ranges from 0 (non-oral feeding) to 100 (unrestricted diet); understandability of speech (UOS) subscale measures the degree a clinician is able to understand the participant's speech, subscale ranges from 0 (never understandable) to 100 (always understandable); eating in public (EIP) subscale, rating based on the participant's response to the questions of whom he/she eats with and in what setting, subscale ranges from 0 (always eats alone) to 100 (no restriction of place, food, or companion). Change from baseline: negative value represents a decrease in function and a positive value represents an increase in function.
Time Frame: Baseline, Day 1 of Cycles 2, 4, 6, cetuximab monotherapy Cycles 2 and 4 (21-day cycle)
Population: All treated participants who had PSS-HNC assessments at baseline and in Cycles 2, 4, 6, cetuximab monotherapy Cycles 2 and 4. Exclude those from a noncompliant study site.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cetuximab + Pemetrexed + Carboplatin/Cisplatin
Number analyzed (Participants) | 52
units on a scale
  Change in NOD at Cycle 2 (n=52) | 4.62 (18.63)
  Change in UOS at Cycle 2 (n=52) | -2.40 (18.69)
  change in EIP at Cycle 2 (n=52) | 2.88 (21.38)
  Change in NOD at Cycle 4 (n=34) | 3.24 (24.58)
  Change in UOS at Cycle 4 (n=35) | -0.71 (19.63)
  Change in EIP at Cycle 4 (n=34) | -6.62 (24.08)
  Change in NOD at Cycle 6 (n=28) | 9.29 (24.78)
  Change in UOS at Cycle 6 (n=28) | -1.79 (16.57)
  Change in EIP at Cycle 6 (n=28) | -1.79 (28.81)
  Change in NOD at monotherapy Cycle 2 (n=16) | 11.88 (32.29)
  Change in UOS at monotherapy Cycle 2 (n=16) | -4.69 (16.38)
  Change in EIP at monotherapy Cycle 2 (n=17) | -4.41 (35.61)
  Change in NOD at monotherapy Cycle 4 (n=9) | 8.89 (18.33)
  Change in UOS at monotherapy Cycle 4 (n=9) | 2.78 (23.20)
  Change in EIP at monotherapy Cycle 4 (n=9) | 2.78 (23.20)

6. Other Pre Specified Outcome: Number of Participants Who Died While on Treatment and Died During 30-Day Post-Treatment Discontinuation Follow-Up (FU)
Description: Presented are the number of participants who died due to adverse events (AEs) while on treatment and participants who died due to progressive disease (PD) during the 30-day post-treatment discontinuation FU.
Time Frame: From enrollment to 30 days post-treatment discontinuation up to 26.4 months
Population: All enrolled participants who received at least 1 dose of any study drug.
Measure: Number; unit: participants
Arm/Group | Cetuximab + Pemetrexed + Carboplatin/Cisplatin
Number analyzed (Participants) | 69
participants
  Due to AE while on treatment | 3
  Due to PD during 30-day FU | 5

ADVERSE EVENTS:
Groups:
- Cetuximab + Pemetrexed + Carboplatin: Cetuximab loading dose of 400 mg/m² administered intravenously on Day 1 of Cycle 1; subsequently 250 mg/m² administered intravenously weekly.
  Pemetrexed 500 mg/m² administered intravenously on Day 1 of every 21-day cycle, 1 hour after cetuximab.
  Carboplatin AUC 5 administered intravenously on Day 1 of every 21-day cycle, 30 minutes after pemetrexed.
  Maximum 6 cycles. Participants who did not experience disease progression after 6 cycles continued on cetuximab (250 mg/m² intravenously weekly) monotherapy until disease progression.
- Cetuximab + Pemetrexed + Cisplatin: Cetuximab loading dose of 400 mg/m² administered intravenously on Day 1 of Cycle 1; subsequently 250 mg/m² administered intravenously weekly.
  Pemetrexed 500 mg/m² administered intravenously on Day 1 of every 21-day cycle, 1 hour after cetuximab.
  Cisplatin 75 mg/m² administered intravenously on Day 1 of every 21-day cycle, 30 minutes after pemetrexed.
  Maximum 6 cycles. Participants who did not experience disease progression after 6 cycles continued on cetuximab (250 mg/m² intravenously weekly) monotherapy until disease progression.
Arm/Group | Cetuximab + Pemetrexed + Carboplatin | Cetuximab + Pemetrexed + Cisplatin
Serious Adverse Events (participants affected / at risk) | 23/63 | 3/6
Other Adverse Events (participants affected / at risk) | 63/63 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cetuximab + Pemetrexed + Carboplatin (N=63) | Cetuximab + Pemetrexed + Cisplatin (N=6)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Haemorrhagic disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (3) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Face oedema (General disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (2) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (2) | 0 (0)
Lung abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Arterial rupture (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cetuximab + Pemetrexed + Carboplatin (N=63) | Cetuximab + Pemetrexed + Cisplatin (N=6)
Anaemia (Blood and lymphatic system disorders) | 40 (60) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 8 (8) | 1 (4)
Neutropenia (Blood and lymphatic system disorders) | 22 (33) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 31 (58) | 3 (6)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Dry eye (Eye disorders) | 2 (2) | 1 (1)
Growth of eyelashes (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 6 (6) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 6 (6) | 1 (1)
Constipation (Gastrointestinal disorders) | 24 (29) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 17 (22) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 7 (7) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 6 (7) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 (6) | 0 (0)
Lip ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 24 (33) | 5 (6)
Salivary hypersecretion (Gastrointestinal disorders) | 2 (2) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 10 (12) | 2 (2)
Vomiting (Gastrointestinal disorders) | 10 (11) | 4 (6)
Asthenia (General disorders) | 8 (8) | 1 (1)
Catheter site erythema (General disorders) | 1 (1) | 1 (1)
Catheter site inflammation (General disorders) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 1 (1) | 1 (1)
Chills (General disorders) | 5 (5) | 0 (0)
Face oedema (General disorders) | 3 (4) | 1 (1)
Facial pain (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 44 (47) | 5 (5)
Inflammatory pain (General disorders) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 22 (30) | 3 (4)
Pain (General disorders) | 8 (10) | 0 (0)
Pyrexia (General disorders) | 12 (13) | 1 (1)
Thrombosis in device (General disorders) | 0 (0) | 1 (1)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Candida infection (Infections and infestations) | 6 (8) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 1 (1)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 1 (2)
Paronychia (Infections and infestations) | 7 (7) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 3 (3)
Ear injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (4) | 1 (1)
Blood magnesium decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 4 (7) | 0 (0)
Platelet count decreased (Investigations) | 5 (8) | 0 (0)
Weight decreased (Investigations) | 9 (9) | 3 (3)
White blood cell count decreased (Investigations) | 10 (19) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 23 (25) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 13 (17) | 4 (6)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (5) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 5 (6) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 13 (14) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 27 (37) | 2 (8)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (6) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 8 (8) | 1 (1)
Dysgeusia (Nervous system disorders) | 5 (5) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 7 (8) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 6 (6) | 1 (1)
Depression (Psychiatric disorders) | 12 (12) | 0 (0)
Insomnia (Psychiatric disorders) | 6 (6) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 2 (3)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 5 (6) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 21 (32) | 4 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 14 (16) | 3 (3)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 5 (6) | 0 (0)
Onycholysis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (7) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 26 (49) | 2 (6)
Skin fissures (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Eyelid operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Gastrostomy (Surgical and medical procedures) | 2 (2) | 1 (2)
Hypotension (Vascular disorders) | 8 (11) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 2 (2) | 1 (1)

LIMITATIONS AND CAVEATS:
Efficacy populations excluded data from a noncompliant site (11 participants).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days